CLINICAL TRIAL: NCT03703193
Title: Dry Needling for Shoulder Pain and Presence of Post-needling Induced-Pain in PAtients Who Had Suffered a Stroke
Brief Title: Dry Needling for Shoulder Pain in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, César Fernández-de-las-Peñas, Director of Department, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: URJC1512201600817
Record Dates: First submitted 2018-10-06; First posted 2018-10-11 (Actual); Last update posted 2018-12-28 (Actual); Status verified 2018-12

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Dry Needling; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling (Experimental): The experimental group will receive a single session of modulatory interventions combined with a single session of dry needling into the shoulder muscles which active trigger points will reproduce the shoulder pain symptoms.
  Interventions: Other: Dry Needling
- Physical Therapy (Active Comparator): This group will receive a single session of modulatory interventions targeting modulation of central nervous system.
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Dry Needling — A single session of modulatory interventions combined with a single session of dry needling into the shoulder muscles which active trigger points will reproduce the shoulder pain symptoms.
  Arms: Dry needling
Other: Physical Therapy — A single session of modulatory interventions targeting modulation of central nervous system.
  Arms: Physical Therapy

SUMMARY:
Spasticity and pain, particularly int he shoulder region, are the most common impairments experienced by subjects who had experienced a stroke. There is preliminary evidence supporting the role of dry needling for spasticity in patients who had suffered from a stroke. Few data exists on the effects on shoulder pain. In addition, it has been shown that application of dry needling induces post-needling soreness in individuals with musculoskeletal pain. No previous study has investigated the presence and the duration of post-needling soreness in individuals who had experienced a stroke.

ELIGIBILITY:
Inclusion Criteria:

* first-ever unilateral stroke;
* hemiplegia resulting from stroke;
* age between 30 and 60 years old;
* presence of hypertonicity in the upper extremity;
* pain symptoms in the shoulder
* active trigger points in the shoulder muscles reproducing the shoulder pain symptoms

Exclusion Criteria:

* recurrent stroke;
* absence of active trigger points in the shoulder muscles reproducing shoulder symptoms
* previous treatment with nerve blocks, motor point injections with neurolytic agents for spasticity at any time;
* previous treatment with botulinum toxin-A in the 6 months prior the study;
* severe cognitive deficits;
* other neurologic diseases,
* underlying complex medical conditions, e.g., heart conditions, unstable hypertension, fracture
* fear to needles;
* any contraindication for deep dry needling, e.g., anticoagulants, infections, bleeding, or psychotic.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
Changes in post-dry needling pain intensity with a numerical pain rate scale before and after the intervention | Baseline, 24 hours (1 day) after and 72 hours (3 days) after treatment the intervention
  A Numerical Pain Rate Scale (NPRS, 0-10) will be used to record post-dry needling soreness in the targeted area

SECONDARY OUTCOMES:
Changes in spontaneous shoulder pain with a numerical pain rate scale before and after the intervention | Baseline, 72 hours (3 days) and 168 hours (7 days) after treatment the intervention
  A Numerical Pain Rate Scale (NPRS, 0-10) will be used to assess spontaneous shoulder pain
Presence of active trigger points in the shoulder musculature | Baseline, 72 hours (3 days) and 168 hours (7 days) after treatment the intervention
  Manual palpation of active trigger points in the shoulder muscles will be conducted

CONTACTS AND LOCATIONS:
Locations (1):
- César Fernández-de-las-Peñas, Alcorcón, Madrid, Spain